CLINICAL TRIAL: NCT05053815
Title: Retrospective Study Assessing the Value of Pharmacogenomic Testing in a Program of All-inclusive Care for the Elderly (PACE) Setting
Brief Title: Pharmacogenomic Testing in a Program of All-inclusive Care for the Elderly (PACE) Setting
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: TRHC-PACE-PGX-2021-001
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Pharmacogenomics; Polypharmacy
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pharmacogenomic Testing — Pharmacogenomic testing is done via buccal swab. As this study is retrospective, data from PGx testing has already been collected as a part of routine care.

SUMMARY:
Tabula Rasa HealthCare (TRHC), doing business as CareKinesis, is the first national pharmacy that provides science-based medication risk identification and mitigation technologies and services. CareKinesis utilizes medication decision support tools and pharmacists certified in geriatrics to provide pharmacy services for various healthcare organizations including PACE organizations.

Program of All-inclusive Care for the Elderly (PACE) is a Medicare-Medicaid program that provides comprehensive medical and supportive services to individuals >55 years of age who are certified by their state as needing nursing home care. As an alternative to institutionalization, PACE helps these individuals live safely in their community. The aim of PACE is to improve overall quality of life in four domains (physical, psychological, social, and spiritual) using a multidisciplinary approach. In the United States, the vast majority of PACE organizations collaborate with one pharmacy to dispense drugs, in addition to other pharmacy services, for their population of participants. Presently, CareKinesis services approximately 140 PACE sites, across the country. As a national PACE pharmacy provider since 2011, CareKinesis focuses on improving medication regimens to reduce medication-related risks while enhancing economic, clinical and humanistic outcomes.

DETAILED DESCRIPTION:
Pharmacist-led pharmacogenomics (PGx) clinical services and medication safety reviews are currently being offered to PACE organizations under the direction of licensed healthcare prescribers by CareKinesis d/b/a Tabula Rasa HealthCare. This project aims to include patients enrolled in the PACE organization who received PGx testing. PGx testing was performed by one of several contracted PGx vendors with TRHC (e.g., Corriel, CQuentia, OneOme) at the time. Upon return from the laboratory, PGx results were integrated into TRHC's proprietary Clinical Decision Support System (Medication Risk Mitigation™ Matrix, CareKinesis, Moorestown, NJ) that guides pharmacists to identify DDIs, DGIs, and DDGIs. As part of this workflow, clinical pharmacists utilized PGx results combined with a comprehensive DDI review (via PGx consult, medication safety review, and/or polypharmacy call) to inform their recommendations to PACE prescribers to address medication problems, including those related to DDIs, DGIs, and/or DDGIs (drug-induced phenoconversion). Upon reviewing the pharmacist's recommendation(s) and based on their clinical assessment, PACE prescribers decided whether to implement the recommended changes. This current study plans to collect data retrospectively from the past six years (2016-2021) on specific PGx test results, genotype-guided and interacting drugs, and recommendations, in order to look for any patterns that may help optimize the process of PGx consultation and/or PGx-guided recommendations, with the ultimate goal of reducing adverse drug events and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient received PGx testing; and
2. Patient enrolled in a PACE organization when PGx test results were returned; and
3. PACE organization contractually received pharmacy services from CareKinesis upon PGx return of results.

Exclusion Criteria:

a) Patient did not receive PGx test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in PACE are 55 years of age and older and are eligible for Medicare and Medicaid.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the value of PGx testing for pharmacogenes and subsequent CDSS-informed, pharmacist-led PGx consultation and its impact on recommendations and prescribing decisions. | 1 year
  Quantitative
Measure PGx-guided interventions on improvement of therapy response. | 1 year
  Quantitative
Measure PGx-guided interventions on improvement of adverse drug events. | 1 year
  Quantitative

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare Precision Pharmacotherapy Research and Development Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No